CLINICAL TRIAL: NCT00890825
Title: Phase II, Double-Blind, Randomised, Placebo-Controlled Study to Assess the Efficacy of AZD6244 in Combination With Docetaxel, Compared With Docetaxel Alone, in 2nd Line Patients With KRAS Mutation Positive Locally Advanced Metastatic NSCLC
Brief Title: AZD6244 in Combination With Docetaxel Versus Docetaxel Alone in KRAS Mutation Positive NSCLC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1532C00016
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer (NSCLC); KRAS mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — AZD 6244; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD6244 + Docetaxel (Active Comparator): AZD6244 75 mg bd + Docetaxel 75 mg/m^2
  Interventions: Drug: AZD6244; Drug: docetaxel
- Placebo + Docetaxel (Placebo Comparator): Placebo + Docetaxel 75 mg/m^2
  Interventions: Drug: docetaxel; Drug: Placebo

INTERVENTIONS:
Drug: AZD6244 — oral capsules, 75mg twice daily
  Other Names: Selumetinib
  Arms: AZD6244 + Docetaxel
Drug: docetaxel — 75mg/m2 iv on day 1 of every 21 day cycle
  Other Names: Taxotere
Drug: Placebo — placebo
  Arms: Placebo + Docetaxel

SUMMARY:
The purpose of this study is to compare the efficacy of AZD6244 in combination with docetaxel versus docetaxel alone in patients with KRAS mutation positive locally advanced or metastatic non small cell lung cancer.

DETAILED DESCRIPTION:
The primary objective of this study was to assess the efficacy in terms of overall survival (OS) of AZD6244 in combination with docetaxel, compared with docetaxel alone, in second-line patients with KRAS mutation-positive locally advanced or metastatic NSCLC. Amendment 4 of the CSP altered the primary objective and outcome variable from progression-free survival (PFS) to OS, and the secondary outcome variable changed from OS to PFS.

The secondary objectives of the study were:

* To further assess the efficacy of AZD6244 in combination with docetaxel, compared with docetaxel alone, in second-line patients with KRAS mutation-positive locally advanced or metastatic NSCLC
* To assess the safety and tolerability profile of AZD6244 in combination with docetaxel
* To investigate the use of plasma and serum as a potential source of circulating free tumour DNA (cfDNA) for the analysis of KRAS mutation status
* To investigate the PK of AZD6244 and N-desmethyl AZD6244 and any other known metabolites when AZD6244 is administered in combination with docetaxel.

The exploratory objectives of the study were:

* To assess the prevalence, severity and change over time of advanced NSCLC cancer specific symptoms in patients receiving AZD6244 in combination with docetaxel and docetaxel alone
* To explore potential biomarkers in residual tumour, plasma and/or serum taken for KRAS mutational analysis which may influence development of NSCLC (and associated clinical characteristics) and/or response (optional)
* To investigate the relationship between AZD6244 and/or N-desmethyl AZD6244 and any other known metabolite plasma concentrations or exposure and clinical outcomes, efficacy, AEs, and/or safety parameters if deemed appropriate
* To collect and store deoxyribonucleic acid (DNA), derived from a blood sample, for future exploratory research into genes that may influence response, eg, distribution, safety, tolerability, and efficacy of AZD6244 and/or agents used in combination and/or as comparators (optional).

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic non small cell lung cancer (IIIB-IV)
* Failure of first line anti-cancer therapy (either radiological documentation of disease progression or due to toxicity) in advanced disease or subsequent relapse of disease following first line therapy
* Tumour sample confirmed as KRAS mutation positive (Note: Sample must be available upon enrolment to ship to AZ appointed central laboratory, or mutation status confirmed locally at AstraZeneca agreed local laboratory using agreed methodology, or mutation status confirmed by an accredited (eg CLIA certified) commercial laboratory (eg Genzyme or Lab 21).

Exclusion Criteria:

* Received >1 prior anti-cancer therapy for advanced or metastatic non small cell lung cancer (excluding radiotherapy)
* Prior treatment with a MEK inhibitor or any docetaxel containing regimen (prior treatment with paclitaxel is acceptable)
* Having received an investigational drug within 30 days of starting treatment, or have not recovered from side effects of an investigational drug
* Brain metastases or spinal cord compression unless asymptomatic, treated and stable off steroids and anti-convulsants for at least 1 month

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-04-20 (Actual); Primary Completion 2011-05-11 (Actual); Study Completion 2016-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pasi Janne, Principal Investigator — Dana-Farber Cancer Institute, Boston, USA; Dr. Gabriella Mariani, Study Director — AstraZeneca, Hertfordshire, UK
Locations (51):
- United States (4):
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Boston, Massachusetts
  - Research Site, Columbus, Ohio
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (6):
  - Research Site, Belo Horizonte
  - Research Site, Ijuí
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São Paulo
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (3):
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
- Czechia (3):
  - Research Site, Ostrava
  - Research Site, Prague
  - Research Site, Znojmo
- France (6):
  - Research Site, Brest
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Rennes
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Mosdós
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
- Italy (7):
  - Research Site, Bologna
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Perugia
  - Research Site, Roma
  - Research Site, Rozzano
- Mexico (3):
  - Research Site, México
  - Research Site, Morelia
  - Research Site, Zacatecas City
- Research Site, Lima, Peru
- Spain (5):
  - Research Site, A Coruña
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga

REFERENCES:
- [Derived] Janne PA, Smith I, McWalter G, Mann H, Dougherty B, Walker J, Orr MC, Hodgson DR, Shaw AT, Pereira JR, Jeannin G, Vansteenkiste J, Barrios CH, Franke FA, Crino L, Smith P. Impact of KRAS codon subtypes from a randomised phase II trial of selumetinib plus docetaxel in KRAS mutant advanced non-small-cell lung cancer. Br J Cancer. 2015 Jul 14;113(2):199-203. doi: 10.1038/bjc.2015.215. Epub 2015 Jun 30. PMID 26125448
- [Derived] Janne PA, Shaw AT, Pereira JR, Jeannin G, Vansteenkiste J, Barrios C, Franke FA, Grinsted L, Zazulina V, Smith P, Smith I, Crino L. Selumetinib plus docetaxel for KRAS-mutant advanced non-small-cell lung cancer: a randomised, multicentre, placebo-controlled, phase 2 study. Lancet Oncol. 2013 Jan;14(1):38-47. doi: 10.1016/S1470-2045(12)70489-8. Epub 2012 Nov 28. PMID 23200175
- See also: Cancer Study Locator (For US and Canada sites only) — https://cancerstudylocator.com/azo/home

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Selection of patients was in 2nd line patients with KRAS mutation positive locally advanced or metastatic NSCLC (Stage IIIB - IV).First patient enrolled: 20 April 2009.Last patient last visit: 30 June 2010.Data Cut Off (DCO): 01 May 2011
Period: Overall Study
Arm/Group | AZD6244 + Docetaxel | Placebo + Docetaxel
Started | 44 | 43 (A patient randomized to this arm was excluded from the safety population for not receiving treatment)
Completed | 30 | 29
Not Completed | 14 | 14
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Alive at data cut off (DCO) | 13 | 14

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD6244 + Docetaxel | Placebo + Docetaxel | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (9.22) | 58.6 (8.38) | 58.4 (8.77)
Age, Customized [Count of Participants; unit: Participants]
  Age group : <=55 years | 15 | 15 | 30
  Age group : >55 years | 29 | 28 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 21 | 20 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 41 | 40 | 81
  Black or African American | 1 | 1 | 2
  Other | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 17
  Not Hispanic or Latino | 37 | 33 | 70

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: OS was calculated as the interval from the date of randomisation to the date of patient death (any cause). Patients who had not died at the time of the final analysis, or who withdrew consent, were censored at the last date the patient was known to be alive.
Time Frame: At least 12 months since start of treatment.
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | AZD6244 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 43 | 40
Participants
  Died | 29 | 27
  Alive at DCO | 13 | 13
  Withdrawn | 1 | 0
Statistical Analysis 1: Comparison: AZD6244 + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.2069, Regression, Cox — One-sided p-value. The p-value is associated with the point estimate (e.g. HR comparing AZD6244 + Docetaxel vs Placebo + Docetaxel) on the outcome measure - Overall survival; Analysis adjusted for the following covariates; WHO PS, gender, histology and smoking status; Hazard Ratio (HR) = 0.80, 80% CI 2-sided [0.56 to 1.14] — A Hazard Ratio less than 1 favoured AZD6244 + Docetaxel

2. Secondary Outcome: Progression Free Survival
Description: PFS was defined as the interval between the date of randomisation and the earlier date of objective disease progression per RECIST criteria or death due to any cause in the absence of progression. Patients who did not progress or die at the time of analysis were censored at the time of their latest evaluable objective tumour assessment. This also included patients who withdrew consent.
Time Frame: At least 12 months after start of treatment
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | AZD6244 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 43 | 40
Participants
  Progression | 35 | 36
  Prog. after >2 missed or non-eval. assessments | 1 | 2
  No progression | 7 | 2
Statistical Analysis 1: Comparison: AZD6244 + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.0138, Regression, Cox — One-sided p-value. The p-value is associated with the point estimate (e.g. HR comparing AZD6244 + Docetaxel vs Placebo + Docetaxel) on the outcome measure; The model allowed for the effect of treatment and included terms for WHO PS, gender, histology, and smoking status; Hazard Ratio (HR) = 0.58, 80% CI 2-sided [0.42 to 0.79] — A Hazard Ratio (HR) < 1 favoured AZD6244 + Docetaxel

3. Secondary Outcome: Objective Response Rate
Description: ORR is defined as the ratio of proportions, patients with at least one visit response of CR or PR in AZD6244 + Docetaxel vs Placebo + Docetaxel.
Time Frame: At least 12 months after start of treatment
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | AZD6244 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 43 | 40
Participants
  Response | 16 | 0
  No response | 27 | 40
Statistical Analysis 1: Comparison: AZD6244 + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Two-sided P-value; Odds Ratio (OR) = 37.2, 95% CI 2-sided [23 to 53]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression, the end of response should coincide with the date of progression or death from any cause used for the PFS endpoint.
Time Frame: At least 12 months after start of treatment
Population: MITT
Measure: Mean (Standard Error); unit: Days
Arm/Group | AZD6244 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 43 | 40
Days | 193.4 (0.207) | NA (NA) — No instance of complete or partial response was recorded for this arm.

5. Secondary Outcome: Change From Baseline in Tumour Size at 6 Week.
Description: Percentage change from baseline in tumour size at 6 week. Values calculated as tumour sizes at 6 weeks minus value at baseline.
Time Frame: 6 weeks after first dose of treatment
Population: MITT
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage change from baseline
Arm/Group | AZD6244 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 43 | 40
Percentage change from baseline | -16.98 [-27.1 to -6.85] | 0.05 [-9.84 to 9.93]
Statistical Analysis 1: Comparison: AZD6244 + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.004, ANCOVA — One-sided p-value. The p-value is associated with the point estimate comparing AZD6244 + Docetaxel vs Placebo + Docetaxel on the outcome measure; LS means were adjusted for baseline tumour size, time from baseline scan to randomisation, WHO PS, gender, histology, and smoking status; LSmeans difference = -17.03, 80% CI 2-sided [-25.2 to -8.86] — (AZD6244 + Docetaxel) - (Placebo + Docetaxel)

6. Secondary Outcome: Change From Baseline in Tumour Size at Week 12
Description: Percentage change from baseline in tumour size at Week 12. Values calculated as tumour sizes at 12 weeks minus value at baseline.
Time Frame: 12 weeks
Population: MITT
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change from baseline
Arm/Group | AZD6244 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 43 | 40
Percent change from baseline | -19.38 [-34.7 to -4.09] | 6.62 [-8.31 to 21.54]
Statistical Analysis 1: Comparison: AZD6244 + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -26.0, 80% CI 2-sided [-38.34 to -13.7] — (AZD6244 + Docetaxel) - (Placebo + Docetaxel)

7. Secondary Outcome: Alive and Progression-Free at 6 Months
Description: Percentage of patients alive and progression-free at 6 months
Time Frame: 6 months after first dose of treatment
Population: MITT
Measure: Number; unit: percentage
Arm/Group | AZD6244 + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 43 | 40
percentage | 37.1 | 15.8
Statistical Analysis 1: Comparison: AZD6244 + Docetaxel vs Placebo + Docetaxel; Test type: Superiority or Other; p = 0.0158, Log Rank — [p-value comment as in outcome 2, analysis 1]; Confidence interval (CI) used Greenwood's formula for the standard error of a survival estimate; Hazard Ratio (HR) = 0.54, 80% CI 2-sided [0.37 to 0.78] — A hazard ratio (HR) <1 favours AZD6244 75 mg bd+Docetaxel

ADVERSE EVENTS:
Time Frame: Over a minimum period of 12 months since start of treatment, or the date of the final analysis of the data, whichever is the later
Arm/Group | AZD6244 + Docetaxel | Placebo + Docetaxel
Serious Adverse Events (participants affected / at risk) | 26/44 | 13/42
Other Adverse Events (participants affected / at risk) | 43/44 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6244 + Docetaxel (N=44) | Placebo + Docetaxel (N=42)
Febrile neutropena (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Neutropena (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram t wave inversion (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6244 + Docetaxel (N=44) | Placebo + Docetaxel (N=42)
Diarrhoea (Gastrointestinal disorders) | 32 (32) | 7 (7)
Nausea (Gastrointestinal disorders) | 19 (19) | 12 (12)
Vomiting (Gastrointestinal disorders) | 19 (19) | 9 (9)
Stomatitis (Gastrointestinal disorders) | 16 (16) | 8 (8)
Constipation (Gastrointestinal disorders) | 14 (14) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 8 (8) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 1 (1)
Fatigue (General disorders) | 12 (12) | 14 (14)
Asthenia (General disorders) | 31 (31) | 28 (28)
Oedema peripheral (General disorders) | 18 (18) | 7 (7)
Pyrexia (General disorders) | 12 (12) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (8)
Dysonoea exertional (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (13) | 9 (9)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 17 (17) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 17 (17) | 15 (15)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 15 (15) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Headache (Nervous system disorders) | 6 (6) | 5 (5)
Dysgeusia (Nervous system disorders) | 5 (5) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 5 (5) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Vision blurred (Eye disorders) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less